CLINICAL TRIAL: NCT05735600
Title: Leveraging Cultural Health Beliefs and Actions to Improve Latinx Family Wellness
Brief Title: Latinx Family Wellness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding/financial issues
Sponsor: Ana Maria Linares (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Ana Maria Linares, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 77822
Record Dates: First submitted 2023-01-10; First posted 2023-02-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; Latinx; Intervention; Deep level education
MeSH Terms: conditions — Pediatric Obesity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two complementary theoretical frameworks inform the proposed study. Social-Ecological Framework suggests that families are nested within multiple social contexts that can influence children's weight. At the macro level, policies can shape child obesity by supplementing families' ability to afford food (e.g., food stamps, income supports), at the messo (community) level, the built and social environments influence child obesity by providing or inhibiting access to healthy food options and safe areas to engage in physical activity. Within the family domain, family attributes, behaviors, functioning, and parental factors, directly shape child obesity. AyUDA targets the family domain by centering obesogenic (obesity-promoting) aspects and mechanisms within families. In concert with this domain, investigators draw from Social Learning Theory to account for how to influence change within the family domain by targeting parenting attitudes and behaviors.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization occurs after the baseline interview. The investigators will prepare ordered envelopes that contain the treatment assignments, one set for each stratum. Within each stratum, the treatment assignments will be placed in blocks of 10 (i.e., five assignments for each of the treatment conditions). Participants will be informed in the assigned group without mentioning if it's the intervention or match control group. Data will be collected by the trained RS who are blind to the study conditions of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual (Experimental): This group will participate in weekly virtual group sessions facilitated by a culturally similar and trained health educator (Promotora). The virtual modules will be on a platform such as Zoom and will last approximately 90 minutes each. Each module will last 60 minutes with the following three components: 1) 15-minute video on behavior change-related module objective, 2) 15-minute vignette/story depicting a family implementing behavior change, and 3) 15-minute discussion on creating goals and overcoming barriers for behavior change pertaining to the module. The remaining 15-minutes will ask participants to share what worked well towards achieving goals set in the prior module
  Interventions: Behavioral: AyuDa Virtual: Aprender y Utilizar Decisiones Apreciables (Spanish) - Learning and Utilizing Significant Choices (English)
- Traditional (Active Comparator): This group will get the same educational materials in writing (slides with information from video, written story, and instructions on goal setting and overcoming barriers) and receive a phone call from one of the researchers each week (5 weeks in a row) to provide an opportunity to respond questions, comments, and provide guidance about following the recommendations of the written material
  Interventions: Behavioral: AyuDa Written: Aprender y Utilizar Decisiones Apreciables (Spanish) - Learning and Utilizing Significant Choices (English)

INTERVENTIONS:
Behavioral: AyuDa Virtual: Aprender y Utilizar Decisiones Apreciables (Spanish) - Learning and Utilizing Significant Choices (English) — The intervention was developed based on the Social Learning Theory, considering both environmental and cognitive factors influencing parent behavior and modeling for children. Researchers have modified a five-module virtual intervention from the "Cooking Healthy and Delicious Manual (Cocinando Delicioso y Saludable Manual, Spanish version), which incorporates behavior change strategies for improving diet quality, screen time, physical activity/sedentary behavior, socioeconomic status/food security, and sleep duration.
  Arms: Virtual
Behavioral: AyuDa Written: Aprender y Utilizar Decisiones Apreciables (Spanish) - Learning and Utilizing Significant Choices (English) — The intervention was developed based on the Social Learning Theory, considering both environmental and cognitive factors influencing parent behavior and modeling for children. Researchers have modified a five-module virtual intervention from the "Cooking Healthy and Delicious Manual (Cocinando Delicioso y Saludable Manual, Spanish version), which incorporates behavior change strategies for improving diet quality, screen time, physical activity/sedentary behavior, socioeconomic status/food security, and sleep duration.
  Arms: Traditional

SUMMARY:
Childhood is an opportune time to intervene in obesity because behaviors that are developed during this time can have long-lasting effects and disrupt trajectories of obesity. This proposal aims to test the feasibility (i.e., participant acceptance, adherence, and retention) of a family-oriented intervention "AyUDA" (Aprender y Utilizar Decisiones Apreciables-Learning and Utilizing Significant Choices). The culturally tailored, two-arm adapted intervention to engage Latinx parents in healthy feeding and lifestyle practices for their children 2-5 years old, thereby reducing early childhood overweight and obesity. The investigators will use concepts of the Social-Ecological Framework for Obesity among Latinx, and the Social Learning Theory that emphasizes the importance of observing, modeling, and imitating behaviors. This approach includes a community engagement partnership with one clinic that serves a great number of Latinx families with 2-5 aged children in Central Kentucky (General Pediatric Clinic-Clinica Amiga). The investigators propose a two-arm randomized clinical trial (RCT) randomly assigning participants to either a telehealth deep cultural level group or a culturally traditional educational group in a sample of 40 Latinx families who will be followed for six months after the intervention. Moreover, investigators will explore short-term changes of the intervention on dietary behavior changes and anthropometric measurements among family members. The feasibility study will inform effect sizes that will be used to estimate statistical power for a future R01 on Community Level Interventions to Improve Minority Health and Reduce Health Disparities, National Institute of Health (NIH).

DETAILED DESCRIPTION:
The feasibility and effectiveness of a family-oriented intervention entitled "AyUDA" will be tested. The AyUDA intervention will provide Latinx families with culturally tailored modules to take control of modifiable behaviors and help them avoid obesogenic behaviors. This study has a longitudinal RCT study design. The study will be conducted in the University of Kentucky Friendly Clinic (Clinica Amiga). Participants will be followed for six months after the intervention. At least one adult who agrees to participate will sign the informed consent and HIPAA authorization, including the children's assent form. We anticipate that recruitment would include non-English speaking subjects due to Latinx self-identity, and for this reason, consent will be obtained in Spanish. The PIs, Co-I, and RP are fluent in English/Spanish and familiar with Latinx culture. Randomization: Randomization occurs after the baseline interview. Researchers will prepare ordered envelopes that contain the treatment assignments, one set for each stratum. Within each stratum, the treatment assignments will be placed in blocks of 10 (i.e., five assignments to each of the treatment conditions). To minimize attrition, complete contact information from participants will be collected and they will be asked to provide the phone number of two individuals who will know how to contact them in the future. Escalating incentives will be provided during data collection encounters to maximize retention. Reminders will be sent monthly for the duration of the study. Data Collection: Data will be collected by the trained RS who are blind to the study conditions at the following times: T1-baseline at recruitment-pre-intervention and randomization, T2-two weeks after the intervention, T3-Three months after the intervention, and T4-Six months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Latinx family of Mexican or Central American descent
* At least one parent 18 years or older; with a child between 2-5 years old and classified as overweight or obese
* Intention to remain in Central Kentucky for at least a year after recruitment
* Access to the internet.

Exclusion Criteria:

* n/a

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Change in scores of the Child Feeding Questionnaire | Baseline and at 1, 3, and 6 months.
  Evaluate change in scores of the Child Feeding Questionnaire (CFQ). A 31-item self-report questionnaire measuring parental beliefs, attitudes, and practices in relation to child feeding. Each item is measured using a 5-point Likert-type scale, with responses across seven factor-based domains. Scores range from 1 to 5 with higher scores indicating higher levels of each domain.
Change in scores of the Caregiver's Feeding Style Questionnaire | Baseline and at 1, 3, and 6 months.
  Evaluate change in scores of the Caregiver's Feeding Style Questionnaire (CFSQ). The CFSQ is a 19-item measure which classifies caregivers into 1 of 4 feeding styles. Items are scored on a 5-point scale (1=never-5=always), with higher scores indicating higher frequency of engagement in a specific feeding style.
Recruitment for AyUDA | From study start until enrollment closes up to 9 months.
  Percentage of eligible participants enrolled during the planned recruitment period.
Intervention completion for AyUDA. | From enrollment to end of intervention at 6 weeks
  Percentage of treatment group participants that complete all intervention sessions
Retention for AyUDA. | From enrollment to end of study at 8 months
  Percentage of participants retained in the study until the conclusion

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and at 6 months after the intervention.
  Evaluation of weight (kilograms) and height (meters) to calculate BMI (kg/m^2) by age and sex following the World Health Organization (WHO) Body mass index percentile by age and sex 2-5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Linares, DNS, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Clinica Amiga, UK Primary Care Pediatrics, Kentucky Clinic South, Lexington, Kentucky
  - Polk Dalton Clinic, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
We plan to make IPD available upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: At the end of the protocol. Approximately December 2024.
Access Criteria: Upon request

REFERENCES:
- [Background] Williams JE, Kabukuru A, Mayo R, Griffin SF. Commentary: A social-ecological perspective on obesity among Latinos. Ethn Dis. 2011 Autumn;21(4):467-72. PMID 22428352
- [Background] Skinner AC, Ravanbakht SN, Skelton JA, Perrin EM, Armstrong SC. Prevalence of Obesity and Severe Obesity in US Children, 1999-2016. Pediatrics. 2018 Mar;141(3):e20173459. doi: 10.1542/peds.2017-3459. PMID 29483202
- [Background] Isong IA, Rao SR, Bind MA, Avendano M, Kawachi I, Richmond TK. Racial and Ethnic Disparities in Early Childhood Obesity. Pediatrics. 2018 Jan;141(1):e20170865. doi: 10.1542/peds.2017-0865. PMID 29269386
- [Background] Beck AL, Hoeft KS, Takayama JI, Barker JC. Beliefs and practices regarding solid food introduction among Latino parents in Northern California. Appetite. 2018 Jan 1;120:381-387. doi: 10.1016/j.appet.2017.09.023. Epub 2017 Sep 23. PMID 28951238